CLINICAL TRIAL: NCT04611529
Title: A Randomized Study of Topical Diclofenac Versus Oral Ibuprofen for Acute Non-radicular Low Back Pain
Brief Title: Acute Low Back Pain. Topical Diclofenac and Oral Ibuprofen.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020-12418
Record Dates: First submitted 2020-10-28; First posted 2020-11-02 (Actual); Results first posted 2024-10-09 (Actual); Last update posted 2024-10-09 (Actual); Status verified 2024-10

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Ibuprofen; Diclofenac

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Oral ibuprofen + topical diclofenac (Experimental): Oral ibuprofen 400mg Topical diclofenac 4gm
  Interventions: Drug: Ibuprofen 400 mg; Drug: Topical diclofenac
- Oral ibuprofen + topical placebo (Active Comparator): Oral ibuprofen 400mg Topical placebo
  Interventions: Drug: Ibuprofen 400 mg
- Oral placebo + topical diclofenac (Active Comparator): Oral placebo Topical diclofenac 4gm
  Interventions: Drug: Topical diclofenac

INTERVENTIONS:
Drug: Ibuprofen 400 mg — Ibuprofen 400mg
  Arms: Oral ibuprofen + topical diclofenac; Oral ibuprofen + topical placebo
Drug: Topical diclofenac — Diclofenac 1% gel 4gm
  Arms: Oral ibuprofen + topical diclofenac; Oral placebo + topical diclofenac

SUMMARY:
This is a randomized, double-blind placebo-controlled study comparing two different treatments for acute low back pain: oral ibuprofen and topical diclofenac. Participants will be randomized to one of three study arms: 1) Oral ibuprofen + topical diclofenac; 2) Oral ibuprofen + topical placebo; 3) Oral placebo + topical diclofenac. Outcomes will be determined at 48 hours (2 days) and 7 days later.

ELIGIBILITY:
Inclusion Criteria:

* Present to Emergency Department (ED) primary for management of Low Back Pain (LBP), defined as pain originating between the lower border of the scapulae and the upper gluteal folds. Flank pain, that is pain originating from tissues lateral to the paraspinal muscles, will not be included.
* Musculoskeletal etiology of low back. Patients with non-musculoskeletal etiologies such as urinary tract infection, ovarian cysts, or influenza like illness will be excluded. The primary clinical diagnosis, at the conclusion of the ED visit, must be a diagnosis consistent with non-traumatic, non-radicular, musculoskeletal LBP.
* Patient is to be discharged home.
* Age 18-69. Enrollment will be limited to adults younger than 70 years because of the increased risk of adverse medication effects in the elderly.
* Non-radicular pain. Patients will be excluded if the pain radiates below the gluteal folds in a radicular pattern.
* Pain duration <2 weeks (336 hours).
* Prior to the acute attack of LBP, back pain must occur less frequently than once per month.
* Non-traumatic LBP: no substantial and direct trauma to the back within the previous month
* Functionally impairing back pain: A baseline score of > 5 on the Roland-Morris Disability Questionnaire

Exclusion Criteria:

* Not available for follow-up
* Pregnant
* Any analgesic medication use on a daily or near-daily basis
* Allergic to or intolerant of investigational medications
* Open wounds or skin breakdown of the lower back
* Contra-indications to investigational medications: 1) known peptic ulcer disease, chronic dyspepsia, or history of gastrointestinal bleed 2) Severe heart failure (NYHA 2 or worse) 3) Chronic kidney disease (GFR <60ml/min) 4) Current use of anti-coagulants 5) cirrhosis (Child Pugh A or worse) or hepatitis (transaminases 2x the upper limit of normal)

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2021-03-02 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Friedman, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment commenced in March 2021 and concluded in June 2023. The study was conducted in 2 Emergency Departments (EDs) both affiliated with Montefiore Medical Center.
Pre-assignment Details: In total, 3281 patients were screened for participation and 198 were randomized into the study. 1 patient was excluded post-randomization due to missing RMDQ data.
Period: 2-day Follow up
Arm/Group | Oral Ibuprofen + Topical Diclofenac | Oral Ibuprofen + Topical Placebo | Oral Placebo + Topical Diclofenac
Started | 65 | 66 | 66
Completed (Having "Completed" the 2-day follow up entailed having data collected for purposes of the Primary Outcome Measure (primary analysis) which was "Change in Pain Disability - Roland Morris Disability Questionnaire (RMDQ) Score." If data was not collected for this Primary Outcome Measure these participants were considered Lost to follow-up at the 2-day timepoint.) | 60 | 60 | 63
Not Completed | 5 | 6 | 3
Not completed — Lost to Follow-up | 5 | 6 | 3
Period: 7-day Follow up
Arm/Group | Oral Ibuprofen + Topical Diclofenac | Oral Ibuprofen + Topical Placebo | Oral Placebo + Topical Diclofenac
Started | 60 | 60 | 63
Completed | 60 | 60 | 63
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Oral Ibuprofen + Topical Diclofenac | Oral Ibuprofen + Topical Placebo | Oral Placebo + Topical Diclofenac | Total
Number analyzed (Participants) | 65 | 66 | 66 | 197
Age, Continuous [Mean (Standard Deviation); unit: years] | 39 (13) | 37 (13) | 39 (13) | 38 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 34 | 18 | 72
  Male | 45 | 32 | 48 | 125
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race/Ethnicity data was aggregated for this study. 1 participant in the 'Oral Ibuprofen + Topical Diclofenac' arm, 3 participants in the 'Oral Ibuprofen + Topical Placebo' arm, and 2 participants in the 'Oral Placebo + Topical Diclofenac' arm refused to provide demographic data.
  Participants
    Asian | 0 | 0 | 2 | 2
    Black/African-American | 9 | 16 | 19 | 44
    Hispanic/Latino | 51 | 43 | 42 | 136
    White | 3 | 2 | 1 | 6
    Multiracial | 0 | 1 | 0 | 1
    Other | 1 | 1 | 0 | 2
    Refused | 1 | 3 | 2 | 6
Region of Enrollment [Number; unit: participants]
  United States | 65 | 66 | 66 | 197
Roland-Morris Disability Questionnaire (RMDQ) at ED visit [Median (Inter-Quartile Range); unit: score on a scale] — The RMDQ is a 24-item patient-reported outcome measure that assesses the level of disability caused by low back pain (LBP). The RMDQ is scored by adding up the number of items the patient checks or answers with "yes". Each item is worth one point, and the score ranges from 0 to 24, with higher scores indicating greater LBP disability
  score on a scale | 19 [13 to 21] | 19 [14 to 22] | 17 [13 to 22] | 18 [13 to 22]
Duration of Low Back Pain before presentation to ED [Median (Inter-Quartile Range); unit: hours] | 72 [24 to 120] | 48 [24 to 98] | 48 [24 to 96] | 56 [24 to 105]
Patients with Previous Episodes of Low Back Pain [Count of Participants; unit: Participants]
  Never Before | 15 | 24 | 18 | 57
  Few Times Before | 36 | 29 | 37 | 102
  Once a Year | 14 | 12 | 9 | 35
  Once a Month | 0 | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain Disability - Roland Morris Disability Questionnaire (RMDQ) Score
Description: Change in Pain Disability was assessed using the Roland-Morris Disability Questionnaire (RMDQ). The RMDQ is a 24-item self-report 'Yes/no' instrument about how low-back pain affects functional activities. Each question is worth one point so scores can range from 0 (no disability) to 24 (severe disability). Change in RMDQ was measured by calculating: 'Baseline RMDQ score - RMDQ Score at 2-day (48 hour) follow-up' with positive scores being indicative of improvement (less pain disability).
Time Frame: Baseline to 48 hours
Population: 5 participants in the 'Oral ibuprofen + topical diclofenac' group; 6 participants in the 'Oral ibuprofen + topical placebo' group; and 3 participants in the 'Oral placebo + topical diclofenac' group were lost to follow-up (LTFU) prior to the 48 hour assessment timepoints.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Oral Ibuprofen + Topical Diclofenac | Oral Ibuprofen + Topical Placebo | Oral Placebo + Topical Diclofenac
Number analyzed (Participants) | 60 | 60 | 63
score on a scale | 8.7 [6.3 to 11.1] | 10.1 [7.5 to 12.7] | 6.4 [4.0 to 8.8]

2. Secondary Outcome: Worst Low Back Pain (LBP)
Description: Worst low back was evaluated by asking patients "How would you describe your worst low back pain in the last 24 hours?" Patients were asked to describe their worst LBP using the terms "Severe", "Moderate", "Mild", or "None". Counts of participants reporting each degree of severity over the prior 24 hours are summarized.
Time Frame: 48 hours
Population: 5 participants in the 'Oral ibuprofen + topical diclofenac' group; 6 participants in the 'Oral ibuprofen + topical placebo' group; and 3 participants in the 'Oral placebo and topical diclofenac' group were lost to follow-up prior to the 48 hour assessment timepoints; however, data was able to be collected from 3 LTFU participants in the Ibuprofen + Diclofenac group.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Ibuprofen + Topical Diclofenac | Oral Ibuprofen + Topical Placebo | Oral Placebo + Topical Diclofenac
Number analyzed (Participants) | 63 | 60 | 63
Participants
  None | 5 | 11 | 8
  Mild | 27 | 28 | 21
  Moderate | 18 | 14 | 23
  Severe | 13 | 7 | 11

3. Secondary Outcome: Use of Medication for Low Back Pain (LBP)
Description: Participants were asked "During the last 24 hours, have you taken any medication at all for low back pain?" and asked to respond either "Yes" or "No". Counts of participants using medication during the prior 24 hours are summarized.
Time Frame: 48 hours
Population: 5 participants in the 'Oral ibuprofen + topical diclofenac' group; 6 participants in the 'Oral ibuprofen + topical placebo' group; and 3 participants in the 'Oral placebo and topical diclofenac' group were LTFU prior to 48 hour assessment timepoints; however, data was able to be collected from 3 LTFU participants in the Ibuprofen + Diclofenac group. Data was also not collected from 1 other participant in the 'Diclofenac + Placebo' group.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Ibuprofen + Topical Diclofenac | Oral Ibuprofen + Topical Placebo | Oral Placebo + Topical Diclofenac
Number analyzed (Participants) | 63 | 60 | 62
Participants
  Yes | 54 | 53 | 50
  No | 9 | 7 | 12

4. Secondary Outcome: Frequency of Low Back Pain (LBP)
Description: Frequency of Low Back Pain will be evaluated by asking patients "Over the last 24 hours, how often were you in pain?" Patients will be asked to respond to the frequency of their LBP over the prior 24 hours based on a 5-point Likert scale consisting of "Not at all", "Rarely", "Sometimes", "Usually", or "Always". This question will help determine the burdensomeness of the LBP in the patient's daily life. Counts of participants reporting each frequency will be summarized.
Time Frame: 48 hours
Population: Data regarding Frequency of Low Back Pain was not collected.
Arm/Group | Oral Ibuprofen + Topical Diclofenac | Oral Ibuprofen + Topical Placebo | Oral Placebo + Topical Diclofenac
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Return to Usual Activities
Description: The percentage of patients who were able to return to usual activities following treatment will be quantified by asking patients to provide a binary "Yes" or "No" response to a question of whether they were able to return to day-to-day activities. Results will be summarized by treatment group.
Time Frame: 48 hours
Population: Data related to the percentage of patients who were able to return to usual activities was not collected.
Arm/Group | Oral Ibuprofen + Topical Diclofenac | Oral Ibuprofen + Topical Placebo | Oral Placebo + Topical Diclofenac
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Number of Visits to Any Healthcare Provider
Description: The number of visits to any healthcare provider will be determined by asking patients whether they had any planned or emergent inpatient or outpatient visits to any healthcare provider for any reason during the course of the study. Group mean results will be summarized by treatment group.
Time Frame: 48 hours
Population: Data related to the number of visits to any healthcare provider was not collected.
Arm/Group | Oral Ibuprofen + Topical Diclofenac | Oral Ibuprofen + Topical Placebo | Oral Placebo + Topical Diclofenac
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Treatment Satisfaction
Description: Patient satisfaction with the treatment they received will be assessed by their response to a binary "Yes" or "No" question regarding satisfaction with their treatment. Results will be summarized by treatment group.
Time Frame: 48 hours
Population: Data related to treatment satisfaction was not collected.
Arm/Group | Oral Ibuprofen + Topical Diclofenac | Oral Ibuprofen + Topical Placebo | Oral Placebo + Topical Diclofenac
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: Change in Pain Disability - Roland Morris Disability Questionnaire (RMDQ) Score
Description: Change in Pain Disability was assessed using the Roland-Morris Disability Questionnaire (RMDQ). The RMDQ is a 24-item self-report questionnaire about how low-back pain affects functional activities. Each question is worth one point so scores can range from 0 (no disability) to 24 (severe disability). Change in RMDQ was measured by calculating: 'Baseline RMDQ score - RMDQ Score at 7-day follow-up with positive scores being indicative of improvement (less pain disability).
Time Frame: 7 days
Population: 5 participants in the 'Oral ibuprofen + topical diclofenac' group; 6 participants in the 'Oral ibuprofen + topical placebo' group; and 3 participants in the 'Oral placebo + topical diclofenac' group were lost to follow-up prior to the 7-day assessment timepoints.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Oral Ibuprofen + Topical Diclofenac | Oral Ibuprofen + Topical Placebo | Oral Placebo + Topical Diclofenac
Number analyzed (Participants) | 60 | 60 | 63
score on a scale | 10.7 [8.4 to 13.0] | 12.2 [9.8 to 14.6] | 9.5 [7.1 to 12.0]

9. Secondary Outcome: Worst Low Back Pain (LBP)
Description: as for outcome 2
Time Frame: 7 days
Population: 5 participants in the 'Oral ibuprofen + topical diclofenac' group; 6 participants in the 'Oral ibuprofen + topical placebo' group; and 3 participants in the 'Oral placebo and topical diclofenac' group were lost to follow-up prior to the 7 day assessment timepoints; however data was able to be collected from 1 of the LTFU participants in the 'Ibuprofen + Diclofenac' group. Data was also not collected from 1 other participant in the 'Diclofenac + Placebo' group.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Ibuprofen + Topical Diclofenac | Oral Ibuprofen + Topical Placebo | Oral Placebo + Topical Diclofenac
Number analyzed (Participants) | 61 | 60 | 62
Participants
  None | 20 | 24 | 15
  Mild | 21 | 23 | 24
  Moderate | 13 | 9 | 16
  Severe | 7 | 4 | 7

10. Secondary Outcome: Use of Medication for Low Back Pain (LBP)
Description: as for outcome 3
Time Frame: 7 days
Population: 5 participants in the 'Oral ibuprofen + topical diclofenac' group; 6 participants in the 'Oral ibuprofen + topical placebo' group; and 3 participants in the 'Oral placebo and topical diclofenac' group were lost to follow-up prior to the 7 day assessment timepoints; however data was able to be collected from 1 of the LTFU participants in the 'Ibuprofen + Diclofenac' group.
Measure: Count of Participants; unit: Participants
Arm/Group | Oral Ibuprofen + Topical Diclofenac | Oral Ibuprofen + Topical Placebo | Oral Placebo + Topical Diclofenac
Number analyzed (Participants) | 61 | 60 | 63
Participants
  Yes | 33 | 31 | 35
  No | 28 | 29 | 28

11. Secondary Outcome: Frequency of Low Back Pain
Description: as for outcome 4
Time Frame: 7 days
Population: Data regarding Frequency of Low Back Pain was not collected.
Arm/Group | Oral Ibuprofen + Topical Diclofenac | Oral Ibuprofen + Topical Placebo | Oral Placebo + Topical Diclofenac
Number analyzed (Participants) | 0 | 0 | 0

12. Secondary Outcome: Return to Usual Activities
Description: as for outcome 5
Time Frame: 7 days
Population: Data related to the percentage of patients who were able to return to usual activities was not collected.
Arm/Group | Oral Ibuprofen + Topical Diclofenac | Oral Ibuprofen + Topical Placebo | Oral Placebo + Topical Diclofenac
Number analyzed (Participants) | 0 | 0 | 0

13. Secondary Outcome: Number of Visits to Any Healthcare Provider
Description: as for outcome 6
Time Frame: 7 days
Population: Data related to the number of visits to any healthcare provider was not collected.
Arm/Group | Oral Ibuprofen + Topical Diclofenac | Oral Ibuprofen + Topical Placebo | Oral Placebo + Topical Diclofenac
Number analyzed (Participants) | 0 | 0 | 0

14. Secondary Outcome: Treatment Satisfaction
Description: as for outcome 7
Time Frame: 7 days
Population: Data related to treatment satisfaction was not collected.
Arm/Group | Oral Ibuprofen + Topical Diclofenac | Oral Ibuprofen + Topical Placebo | Oral Placebo + Topical Diclofenac
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From baseline up to 7 days following treatment
Description: Medication-related adverse events were elicited by asking whether the study medications caused any new symptoms.
Arm/Group | Oral Ibuprofen + Topical Diclofenac | Oral Ibuprofen + Topical Placebo | Oral Placebo + Topical Diclofenac
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/60 | 0/63
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60 | 0/63
Other Adverse Events (participants affected / at risk) | 4/60 | 3/60 | 1/63
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oral Ibuprofen + Topical Diclofenac (N=60) | Oral Ibuprofen + Topical Placebo (N=60) | Oral Placebo + Topical Diclofenac (N=63)
Drowsiness (Nervous system disorders) | 0 | 2 | 0
Pruritis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Muscle Cramp (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Chills (General disorders) | 1 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-12-21): https://cdn.clinicaltrials.gov/large-docs/29/NCT04611529/Prot_SAP_000.pdf
  • Informed Consent Form (2022-12-08): https://cdn.clinicaltrials.gov/large-docs/29/NCT04611529/ICF_001.pdf